CLINICAL TRIAL: NCT04993014
Title: Circulating Tumor Cells and Adjuvant Treatment De-escalation After Neoadjuvant Therapy With Trastuzumab and Pertuzumab for HER2 Positive Early Breast Cancer
Brief Title: Circulating Tumor Cells and Treatment De-escalation After Neoadjuvant Therapy for HER2 Positive Breast Cancer
Acronym: HER2Cell
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Marcelle Goldner Cesca, Clinical Oncologist, AC Camargo Cancer Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2861/20
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Breast Neoplasms; HER2-positive Breast Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 cohorts, based on HER2 positivity in CTCs at baseline of neoadjuvant therapy.
  Cohort 1: HER2 positive CTCs: randomization to adjuvant trastuzumab versus trastuzumab + pertuzumab in patients with pathological complete response Cohort 2: HER2 negative/absent CTCs: randomization to adjuvant trastuzumab versus trastuzumab + pertuzumab in patients with pathological complete response
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1, Arm A - trastuzumab (Active Comparator): Adjuvant trastuzumab for patients with HER2 positive CTCs at baseline
  Interventions: Drug: Trastuzumab; Other: Circulating tumor cells
- Cohort 1, Arm B - Trastuzumab + pertuzumab (Experimental): Adjuvant trastuzumab + pertuzumab for patients with HER2 positive CTCs at baseline
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Other: Circulating tumor cells
- Cohort 2, Arm A - trastuzumab (Active Comparator): Adjuvant trastuzumab for patients with HER2 negative/absent CTCs at baseline
  Interventions: Drug: Trastuzumab; Other: Circulating tumor cells
- Cohort 2, Arm B - Trastuzumab + pertuzumab (Experimental): Adjuvant trastuzumab + pertuzumab for patients with HER2 negative/absent CTCs at baseline
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Other: Circulating tumor cells

INTERVENTIONS:
Drug: Pertuzumab — Adjuvant trastuzumab + pertuzumab (arm B of the 2 cohorts: 1: HER2 positive CTCs at baseline and 2: HER2 negative/absent CTCs at baseline)
  Other Names: Perjeta
  Arms: Cohort 1, Arm B - Trastuzumab + pertuzumab; Cohort 2, Arm B - Trastuzumab + pertuzumab
Drug: Trastuzumab — Adjuvant trastuzumab (arm A of the 2 cohorts: 1: HER2 positive CTCs at baseline and 2: HER2 negative/absent CTCs at baseline) Association with pertuzumab in arm B of the 2 cohorts
  Other Names: Zedora
Other: Circulating tumor cells — Blood sample collection for examination of CTCs at baseline of neoadjuvant therapy. Tests for HER2 positivity will be done.
  Other Names: CTCs

SUMMARY:
Phase II unicentric randomized trial which will include early HER2 positive breast cancer patients, candidate to neoadjuvant therapy with trastuzumab and pertuzumab. Circulating tumor cells will be collected at neoadjuvant therapy baseline.

Patients with pathological complete response will be randomized in 1:1 ratio for adjuvant trastuzumab (arm A) versus trastuzumab + pertuzumab (arm B) in a two factorial design: group A, with HER2 positive CTCs and group B, with HER2 negative/absent CTCs.

DETAILED DESCRIPTION:
Patients with HER2 positive breast cancer (hormone receptors positive or negative), which are candidate to neoadjuvant therapy with pertuzumab and trastuzumab will be included.

Blood samples will be collected at baseline (before neoadjuvant start) for the analysis of CTCs and its positivity for HER2 by IHC and ISH.

Patients with pathological complete response will be included in the randomization phase of the study. There will be 2 cohorts: HER2 positive CTCs at baseline and HER2 negative/absent CTCs at baseline. In each cohort, patients will be randomized in 1:1 ratio for adjuvant trastuzumab versus adjuvant trastuzumab + pertuzumab

ELIGIBILITY:
Inclusion Criteria:

* HER2 positive breast cancer (hormone receptors positive or negative)
* Stage I to III
* Indication for neoadjuvant therapy with chemo (any regimen) + trastuzumab + pertuzumab
* Breast surgery after neoadjuvant therapy
* Preserved coagnition
* ECOG 0-3
* For the randomization phase: pathological complete response (ypT0/ypTis and ypN0)
* Agreement on participation and signature of de ICF

Exclusion Criteria:

* Contradindication for trastuzumab or pertuzumab
* Adjuvant chemotherapy. Hormone therapy is allowed
* Second primary tumor < 5 years, with an exception for treated non-melanoma skin cancer, and in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
HER2 therapy disease-free survival | From adjuvant therapy initiation to recurrence or death by any cause, whichever came first, assessed up to 5 years
  To compare the disease-free survival between trastuzumab and trastuzumab + pertuzumab arms
CTCs disease-free survival | From adjuvant therapy initiation to recurrence or death by any cause, whichever came first, assessed up to 5 years
  To compare the disease-free survival between patients with HER2 positive CTCs at baseline versus HER2 negative/absent CTCs

SECONDARY OUTCOMES:
Prognostic factors for disease-free survival | At baseline and adjuvant therapy (18 months)
Correlation of CTCs and pathological complete response | At baseline
  To evaluate if there is a correlation of HER2 positivity and the number of CTCs/ml and the pathological response
Adverse events | Adjuvant period (1 year)
  To compare the adverse events between trastuzumab and trastuzumab + pertuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle G Cesca, MD, Principal Investigator — A.C. Camargo Cancer Center
Locations (1):
- A.C. Camargo Cancer Center, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No